CLINICAL TRIAL: NCT02481648
Title: A Pilot Study to Evaluate Feasibility of Measuring Exercise's Effects on Molecular Mechanisms of Disease Progression in Newly Diagnosed Prostate Cancer Patients Undergoing Radical Prostatectomy
Brief Title: Feasibility of Measuring Exercise's Effects on Molecular Mechanisms of Disease Progression in Prostate Cancer
Acronym: EMMPC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vancouver Prostate Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EMMPC
Record Dates: First submitted 2015-01-27; First posted 2015-06-25 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM1: Exercise Intervention (Experimental): The exercise program is a 4-12 weeks progressive combined resistance and aerobic exercise for participants from time of diagnosis to RP.
  Participants will undergo twice weekly group-training (four-six participants/group) combined aerobic-resistance sessions (1hr per session), supervised by trained exercise therapists. In addition, participants will undergo home-based aerobic exercise independently three times a week with the goal to meet the current physical activity guidelines for cancer survivors (150min/week of moderate intensity aerobic activity and two resistance training sessions per week). Participants will also be supplied with the Canadian Physical Activity and Sedentary Behavior Guidelines Handbook and accompanying Log Sheets.
  Interventions: Other: Exercise
- ARM2: Control Group (No Intervention): Participants will be asked to exercise as they normally would and will be asked to record their exercise activity on provided activity logs.

INTERVENTIONS:
Other: Exercise
  Arms: ARM1: Exercise Intervention

SUMMARY:
The investigators aim to evaluate the feasibility of a larger clinical trial assessing an exercise program during the "teachable moment" in patients with prostate cancer and measuring its effect on tumor apoptosis signaling, lipogenesis and steroidogenesis. Participants will be randomized between a 4-12 week exercise program or to standard of care only. Participants will be assessed at screening, baseline (day 0), throughout the trial intervention (days 1-84), post-intervention visit (prior to radical prostatectomy) and final study visit 6-months post-radical prostatectomy. At each assessment, physical, biological samples and psychosocial assessments will take place.

ELIGIBILITY:
Inclusion criteria:

* Completed Pre-Screening Consent Form
* Men with CaP, who are deemed suitable by a urologist for RP
* Engaging in <90 minutes/week of moderate-to-vigorous exercise
* BMI <40
* Age >19
* Able to speak and read English (to be able to complete questionnaires)
* Willing to comply with all study procedures (including committing to twice-weekly visits to the study exercise facility and exercise at home) and be available for the duration of the study
* Provide signed and dated informed consent form

Exclusion Criteria:

• Men with a medical, musculoskeletal condition or use of mobility aid that prevents participation in the exercise intervention.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Number of patients screened per month | From start of recruitment to end of recruitment
Feasibility: Number of patients enrolled per month | From start of recruitment to end of recruitment
Feasibility: Proportion of screen eligible patients who enroll | From start of recruitment to end of recruitment
Feasibility: Treatment-specific retention rates | From date of randomization to end of treatment intervention for each participant, an average of 4-12 weeks
Feasibility: Rates of adherence to protocol for the exercise intervention arm and control arm | From date of randomization to end of treatment intervention for each participant, an average of 4-12 weeks
Feasibility: Proportion of planned assessments that are completed respectively | From date of randomization to end of study for each participant, an average of 7 months

SECONDARY OUTCOMES:
Physical Fitness: Godin Leisure-Time Exercise questionnaire (GLTEQ) and activity logs | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of activity at baseline, during the study and at the end of the study
Physical Fitness: Anthropometrics (i.e. BMI & waist circumference) | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of baseline versus end of study anthropometrics
Physical Fitness: Aerobic fitness using a submaximal graded exercise test | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of baseline versus end of study aerobic fitness
Physical Fitness: Functional fitness using the 30-second chair stand and 30-second arm curl | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of baseline versus end of study functional fitness
Physical Fitness: Muscular strength test upper and lower extremity using the 1RM | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of baseline versus end of study muscular strength
Physical Fitness: Blood pressure and pulse | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of baseline versus end of study blood pressure and pulse
Biological: Collection of urine, blood, biopsy and RP specimens | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Ability to collect these samples for each participant will be assessed
Psychosocial: Functional Assessment of Cancer Therapy-Prostate questionnaire (FACT-P) | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of questionnaire scores at baseline versus end of study
Psychosocial: Centre for Epidemiologic Studies Depression scale (CES-D) | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of questionnaire scores at baseline versus end of study
Psychosocial: International Prostate Symptom Score (IPSS) | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of questionnaire scores at baseline versus end of study
Psychosocial: International Index of Erectile Function scale (IIEF) | Baseline (month 0), pre-surgery (4-12 weeks) and 6-months post surgery
  Comparison of questionnaire scores at baseline versus end of study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Black, MD, Principal Investigator — Department of Urologic Sciences, University of British Columbia
Locations (1):
- Vancouver Prostate Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Schulz GB, Locke JA, Campbell KL, Bland KA, Van Patten CL, Black PC, Goldenberg SL, Flannigan R. Taking Advantage of the Teachable Moment at Initial Diagnosis of Prostate Cancer-Results of a Pilot Randomized Controlled Trial of Supervised Exercise Training. Cancer Nurs. 2022 May-Jun 01;45(3):E680-E688. doi: 10.1097/NCC.0000000000001013. Epub 2022 Jan 14. PMID 34608048